CLINICAL TRIAL: NCT05727254
Title: Agility Training for Older Adults: A Randomized Controlled Trial
Brief Title: Agility Training for Older Adults to Improve Fall Risk Factors
Acronym: AgilE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oliver Faude (Other)
Responsible Party: Sponsor-Investigator, Oliver Faude, Prof. Dr., University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2222-00145
Record Dates: First submitted 2023-01-13; First posted 2023-02-14 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Age-Related Loss of Skeletal Muscle Mass; Aging; Sarcopenia; Cognitive Decline
MeSH Terms: conditions — Sarcopenia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with an intervention and a control arm.
Masking Description: Due to the nature of the study (exercise intervention) no masking of participants and intervention providers is possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Agility Training (Experimental): 16 weeks, two times per week, 1 hour of multi-component exercise training, exercise guidelines and exercise diary.
  Interventions: Behavioral: Agility training; Behavioral: Exercise recommendations; Behavioral: Exercise diary
- Control (Active Comparator): Exercise guidelines and exercise diary.
  Interventions: Behavioral: Exercise recommendations; Behavioral: Exercise diary

INTERVENTIONS:
Behavioral: Agility training — Multi-component (strength, balance, cognition) exercise training.
  Arms: Agility Training
Behavioral: Exercise recommendations — Participants are being given the standard recommendations how much exercise and what type older adults should do.
Behavioral: Exercise diary — Participants are instructed to write down their physical activity and exercises.

SUMMARY:
In this randomized controlled trial the effect of 4 months of multi-component (strength, balance, cognition, endurance) exercise training intervention on measures of neuromuscular performance, cognition, and endurance as well as neural adaptations on a central and peripheral level is investigated. 40 subjects are recruited that are generally health and between 60 and 80 years of age. The interventions is based around exercises, where different tasks have to be solved simultaneously rather than serially, as has previously been done.

ELIGIBILITY:
Inclusion Criteria:

* willing to be randomized to either arm
* ability to travel to the sports facility twice a week
* understanding the german language

Exclusion Criteria:

* smoking, obesity
* history of cardiovascular, pulmonary or chronic inflammatory disease
* vision impairments
* orthopaedic problems preventing them from participating in an exercise program
* history of osteoporosis or recent low trauma fracture
* less than two weeks during the intervention period
* not have taken part in a structured exercise program more than once a week in the past three months

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Isometric knee-extension strength | 16 weeks
  Strength in torque (N*m) of the quadriceps femoris muscle. Measured on an isokinetic device in an isometric condition.

SECONDARY OUTCOMES:
Isometric knee-flexion strength | 16 weeks
  Strength in torque (N*m) of the hamstring muscle group measured on an isokinetic device in an isometric condition.
Cognitive Processing Speed | 16 weeks
  Eriksen flanker task performance measured be reaction speed in milliseconds and accuracy in percentage.
Cognitive Impulsiveness | 16 weeks
  Go / No-Go task performance measured by reaction speed in milliseconds and accuracy in percentage.
Balance Performance | 16 weeks
  Staying as stable as possible during ten seconds in tandem stance eyes open condition. Center of pressure sway path length in mm and average sway speed in m/s is calculated.
Hand Grip Strength | 16 weeks
  Using a handheld dynamometer with an extended arm squeezing as hard as possible. Measured in N.
Counter movement jump power | 16 weeks
  Measured on a force plate participants are instructed to jump as high as possible with their hands akimbo. Peak of the time-power curve in Watts.
Blood Pressure | 16 weeks
  Blood pressure cuff on the right arm at the height of the aorta. Measured in mmHG.
Pulse Wave Velocity | 16 weeks
  Estimated from a mobile blood pressure cuff (mobil-O-graph) on the right arm. Measured in m/s.
Retinal vessel diameter | 16 weeks
  A photo is made from the retinal vessels with a static vessel analyzer (camera)through the eye and the vessel diameters are measured in mikrometers.
Quality of Life Questionnaire | 16 weeks
  26 item questionnaire (WHOQOL-Bref). Every answer is rated on a scale from 1 to 5. Aggregate Score from 0 to 100.
Fall Efficacy | 16 weeks
  16 item qestionnaire (Fall Efficacy Scale). Every answer is rated on a scale from 1 to 4.
Sleep Disturbances | 16 weeks
  7 item questionnaire (Insomnia Severity Index). Every answer is rated on a scale from 1 to 5.
Stress | 16 weeks
  10 item qestionnaire (Perceived Stress Scale). Every answer is rated on a scale from 1 to 5.
Depression | 16 weeks
  15 item questionnaire (Center for Epidemiological Studies Depression Scale). Every answer is rated on a scale from 1 to 4.

OTHER OUTCOMES:
Corticospinal Inhibition | 16 weeks
  Difference between paired and single pulse motor evoked potential by transcranial magnetic stimulation.
Voluntary activation | 16 weeks
  Degree of ability to contract the soleus muscle voluntarily.

CONTACTS AND LOCATIONS:
Locations (1):
- Departement für Sport, Bewegung und Gesundheit, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Publication of the raw data along the publication of the results. Data is anonymized. Outcome results of the individual tests are shared.
Supporting Information: Study Protocol, SAP
Time Frame: End of 2023
Access Criteria: Open Access